CLINICAL TRIAL: NCT05837299
Title: A Clinical Study on the Safety and Preliminary Efficacy of IMC008 in the Treatment of CLDN18.2- Positive Advanced Solid Tumors
Brief Title: A Study of IMC008 for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Luo Tianhang, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC008-CT01
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose escalation of 3 dosage groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMC008 dose 1-3 (Experimental): a certain number of IMC008 cell per kg will be infused
  Interventions: Drug: IMC008

INTERVENTIONS:
Drug: IMC008 — allowing 10% dose error
  Other Names: NKG2D receptor-modified autologous CAR -T cells targeting CLDN18.2

SUMMARY:
An open label, multi-center, dose-escalating study to evaluate the safety and preliminary efficacy of IMC008 in CLDN18.2 positive advanced solid tumors.

DETAILED DESCRIPTION:
This study is an open label, multi-center, dose-escalating clinical study to evaluate the safety and preliminary efficacy of IMC008 in the treatment of CLDN18.2 positive advanced solid tumors. DLTs observations will be performed 28 days after IMC008 administration. During the study, regular safety meetings will be held according to the progress of the study, and recommendations will be made on dose escalation, safety of subjects and possible study change.

ELIGIBILITY:
Inclusion Criteria:

* Advanced gastric cancer /esophagogastric junction adenocarcinoma advanced pancreatic cancer.
* Tumor tissue samples of subjects expected to be available with positive for CLDN18.2 immunohistochemistry.
* The expected survival period of the subject is ≥12 weeks.
* The subject needs to have at least one target lesion that can be stably evaluated.
* The ECOG score is 0-1.
* Subject has adequate organ and bone marrow function
* All toxic reactions caused by previous anti-tumor therapy were relieved to grade 0-1.
* Fertility status : Women of childbearing age or men whose sexual partners are women of childbearing age are willing to take medically approved high-efficiency contraceptive measures.
* Subjects must sign and date written informed consent.

Exclusion Criteria:

* Pregnant and lactating women.
* Known history of human immunodeficiency virus infection; acute or chronic active hepatitis B; acute or chronic active hepatitis C. Syphilis antibody positive; Epstein-Barr virus infection; CMV infection.
* Serious infection that is active or poorly controlled clinically.
* Uncontrollable pleural effusion, pericardial effusion, peritoneal effusion existed before enrollment.
* Extensive or diffuse lung metastases or extensive or diffuse liver metastases.
* Oxygen saturation ≤ 95% without oxygen inhalation.
* Suffering from other research diseases that may limit their participation in this study.
* Known past or current hepatic encephalopathy requiring treatment; patients with current or history of central nervous system disease.
* There are heart diseases that need to be treated or hypertension that is poorly controlled by the investigator, poorly controlled after standard treatment type 2 diabetes mellitus.
* Presence of any cardiac clinical symptoms or disorders.
* Evidence of significant coagulopathy or other significant bleeding risk.
* Received systemic steroids equivalent to >15 mg/ day prednisone cumulatively for more than 3 days within 2 weeks prior to apheresis , excluding inhaled steroids.
* Prior or concurrent occurrence of other malignancies, with the following exceptions.
* Subjects who have previously received other gene therapy.
* Allergic/ intolerance to lymphodepletion regimen or CRS treatment drugs or IMC008.
* Subjects with severe mental disorders.
* The investigator assessed the subject's inability or unwillingness to comply with the requirements of the study protocol .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
DLT | within 28 days
  To observe the incidence of dose-limiting toxicity (DLT) after IMC008 infusion

SECONDARY OUTCOMES:
TRAE | up to 96 weeks
  To treatment-related adverse events (TRAE) and severity
PFS | upto 96 weeks
  To evaluate the progression-free survival of IMC008 in patients with CLDN18.2 positive advanced solid tumor
Objective response rate (ORR) | upto 96 weeks
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Tmax | upto 96 weeks
  Tmax of CAR-T cells in the blood.
Lymphocyte subsets | upto 96 weeks
  CAR-T cell lymphocyte subsets/phenotype, etc.
OS | upto 96 weeks
  To evaluate the overall survival of of IMC008 in patients with CLDN18.2 positive advanced solid tumor

CONTACTS AND LOCATIONS:
Overall Officials: Tianhang Luo, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China